CLINICAL TRIAL: NCT02404987
Title: A Prospective, Observational Study, of a High Calorie and Protein Oral Nutritional Supplement, in an Older Malnourished Spanish Population
Brief Title: An Oral Nutritional Supplement Study in Older Malnourished Spanish Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA07
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nutritional Supplement: Free living and residing and nursing home malnourished patients
  Interventions: Other: Nutritional Supplement

INTERVENTIONS:
Other: Nutritional Supplement

SUMMARY:
Post-marketing observational study of a nutritional care plan, including a higher calorie, higher protein oral nutritional supplement (ONS), prescribed to Spanish patients, both free living and residing and nursing homes, who have been identified as malnourished. The objective is to assess the impact of the ONS on body weight, activities of daily living and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to any participation in the study.
* Considered malnourished, or is at risk for malnutrition based on NRS 2002 score ≥3.
* ≥65 years of age.
* Conforms to the requirements set forth on the study product label.
* Under the care of a health care professional for malnutrition and has recently (within the last 7 days prior to participating in this study) been prescribed 2 servings/d of the study ONS, orally, by their health care professional.
* Free living or residing in a nursing home.
* Estimated, or measured, glomerular filtration rate >60ml/min/1.73m2 (Modification of Diet in Renal Disease (MDRD) Study equation) within 60 days of beginning their nutritional care plan.
* Body mass index (BMI) is <30 kg/m2.
* Study physician determines the subject is fit to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Spanish patients, both free living and residing and nursing homes, who have been identified as malnourished.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Change from baseline to 12 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Change from baseline to 12 weeks
  BMI will be calculated: weight (kg)/ height (cm)^2
Katz Activities of Daily Living | Change from baseline to 12 weeks
  A standardized, validated tool that asks about independence in bathing, dressing, toileting, transferring, continence and feeding.
Quality of Life | Change from baseline to 12 weeks
  EQ5D, self-reported quality of life tool

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Sanz Barriuso, RD, PharmD, Study Chair — Abbott Nutrition
Locations (1):
- Hospital Clinico Universitario, Valladolid, Spain